CLINICAL TRIAL: NCT05401643
Title: Evaluación Del Impacto de Una intervención Multidimensional, Con Herramientas TIC, en la Calidad de Vida de Las Pacientes Supervivientes al cáncer de Mama
Brief Title: Evaluation of the Impact of a Multidimensional ICT Intervention on the Quality of Life of Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Fundacion iSYS, internet, salud y sociedad (Unknown)
Responsible Party: Principal Investigator, Imma Grau, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2020/0971
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Breast Neoplasms; Quality of Life; Survivorship
Keywords: Digital Health; mHealth; Quality of Life; Patient Support; eHealth
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, longitudinal, randomized 1:1 trial, with two arms: a control group and an intervention group. The intervention will be 12 months long for each participant. There will be a total of 150 participants. Half (75) will comprise the control group and half (75 more) the intervention group. Only the intervention group will have access to the Xemio mobile app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth intervention (Experimental): Installation of the mHealth application Xemio in the participant's smartphones. Voluntary use of the application for 12 months. Outcome measures collected every 3 months.
  Interventions: Other: Xemio mobile application
- Control (No Intervention): No application installed. Outcome measures collected every 3 months.

INTERVENTIONS:
Other: Xemio mobile application — The study consists in a mHealth intervention provided through the Xemio mobile application for breast cancer survivors. This application is installed in the personal smartphones of the participants after they are randomized in the mHealth intervention group. The Xemio app components are symptom tracking, up-to-date calendar of events organized by patient's organizations, virtual talks with experts, articles regarding new information of the disease, physical activity tracking, and evidence-based information regarding symptoms, non-pharmacological treatments for side effects, and information about common drugs to treat breast cancer. The participants can freely use the Xemio mobile application for a total of 12 months.
  The control group does not have access to the Xemio application for the duration of the study but they are offered access to it at the completion of the intervention. The participants of both arms continued to receive the usual care from their oncology teams.
  Arms: mHealth intervention

SUMMARY:
mACMA is a pilot study that is developed for breast cancer survivors of the Hospital Clinic of Barcelona. The objective of this study is to evaluate the progress in quality of life through the introduction of a mobile phone App that allows for symptom tracking, physical activity tracking and a calendar of patient-oriented events organized by patient organizations. This study is a two-arm randomized clinical trial.

This project has received funding from the European Union's Horizon 2020 research and innovation program under grant agreement No 875351.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnostic of breast cancer
* Free of disease at the time of randomization
* Signed consent form
* Possession of a smartphone and ability to use smartphone applications
* Patients belonging to the ACMA group o being treated at Hospital Clínic
* Without diagnosis of neurodegenerative disorders that prevent participation in the study

Exclusion Criteria:

* Acute process of cancer at the moment of recruitment
* Active treatment for cancer (chemotherapy, radiotherapy)
* Comorbidities such as heart failure NYHA class 4, COPD,...
* Inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life of cancer patients | Baseline, t=3 months, t= 6 months, t= 9 months, t= 12 months (completion of the study)
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30). Measured as 0-100.
Change in Quality of Life specific to breast cancer patients | Baseline, t=3 months, t= 6 months, t= 9 months, t= 12 months (completion of the study)
  European Organisation for Research and Treatment of Cancer Breast 23 (EORTC BR-23). Measured as 0-100.

SECONDARY OUTCOMES:
Change in Anxiety and Depression | Baseline, t=3 months, t= 6 months, t= 9 months, t= 12 months (completion of the study)
  Hospital Anxiety and Depression Scale (HADS). Measured as 0-21, 0 being the best and 21 being the worst.
Change in Loneliness | Baseline, t=3 months, t= 6 months, t= 9 months, t= 12 months (completion of the study)
  Three-Item Loneliness Scale. Measured as 0-9, 0 being the best, 9 being the worst.
Steps | Continuous (12 months)
  Number of steps taken daily by study participants
Change in Weight | Baseline and t= 12 months
  Weight (kg) measured with a bioimpedance scale
Change in Body Mass Index (BMI) | Baseline and t= 12 months
  BMI (kg/m^2) measured with a bioimpedance scale
Change in Fat mass percentage | Baseline and t= 12 months
  Fat mass percentage measured with a bioimpedance scale
Change in muscle mass percentage | Baseline and t= 12 months
  Muscle mass percentage measured with a bioimpedance scale
Change in Social Determinants of Health | Baseline and t= 12 months
  Smoking status, education level, employment status, zip code, alcoholic beverage consumption, civil status
Symptoms reported with the Xemio mobile application | Continuous (12 months)
Use of the Xemio mobile application | Continuous (12 months)
  Time that the Xemio mobile application is open in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Imma Grau, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not shared as it is stated in the approved informed consent and protocol approved by the institution's Ethics Committee. Some of the data collected in this study contains clinical information, hence it is sensible information that needs to remain private.